CLINICAL TRIAL: NCT03360851
Title: DiagNostic Intervention Study of Low-dose CT and multipleX PCR on Antibiotic Treatment and Outcome of Community-Acquired Pneumonia
Brief Title: DiagNostic Study of Low-dose CT and multipleX PCR on Antibiotic Treatment and Outcome of Community-Acquired Pneumonia
Acronym: CAP-NEXT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic has changed routine diagnostic workup of patients admitted with pneumonia. Continuation of the trial was felt to invalidate the study results.
Sponsor: MJM Bonten (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor-Investigator, MJM Bonten, Professor of molecular epidemiology of infectious diseases, head of department of medical microbiology, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61857.041.17
Record Dates: First submitted 2017-10-27; First posted 2017-12-04 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia; low-dose CT; low-dose computed tomography; point of care testing; multiplex PCR; lower respiratory tract infection; antibiotic stewardship
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomised trial with historical control period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Low-dose CT (Experimental): A low-dose chest CT-scan will be performed either directly from the ER or from the medical ward as soon as possible but within 24 hours of admission. The CT will be performed with a radiation dose <0.5 mSv for a 70kg patient, as a replacement or in addition to the chest radiograph. Pregnancy will be an exclusion criterion for CT because of unwanted radiation exposure. CT interpretation will be performed by a radiologist. Test results will be communicated to the treating physician. Recommendations based on the CT may be to discontinue antibiotics in case of a noninfectious diagnosis that explains the presented signs and symptoms and to start treatment for the alternative diagnosis if needed, or to re-evaluate the CAP diagnosis if no signs of lobar or bronchopneumonia are detected on the CT.
  Interventions: Diagnostic Test: low-dose CT
- PoC-PCR (Experimental): The FilmArray real-time multiplex PCR (Biofire; bioMérieux) is a Point-of-Care PCR with a panel of respiratory viruses (adenovirus, coronavirus, human metapneumovirus, human rhinovirus/enterovirus, influenza A and B, parainfluenza virus, and respiratory syncytial virus), and three atypical pathogens (Mycoplasma pneumoniae, Chlamydophila pneumoniae, and Bordetella pertussis), which will be performed on nasopharyngeal swab samples. Test results will be made available to the treating physician immediately. The treatment recommendation could be adaptation of antibiotic treatment for a documented atypical pathogen, a recommendation to not start or discontinue antibiotics when a virus is the only detected pathogen, or a recommendation to discontinue coverage of atypical pathogens.
  Interventions: Diagnostic Test: PoC-PCR
- Standard care (No Intervention): All hospitals will continue the antibiotic stewardship activities employed during the baseline period as part of standard care. A representative of the Antibiotics-team (Team consisting of clinical microbiologists, infectious diseases specialist and clinical pharmacists supervising in-hospital antibiotic use) will monitor the empirical antibiotic treatment of patients hospitalized with CAP to non-ICU wards and provide feedback if indicated.

INTERVENTIONS:
Diagnostic Test: low-dose CT — see arm/group description
  Arms: Low-dose CT
Diagnostic Test: PoC-PCR — see arm/group description
  Arms: PoC-PCR

SUMMARY:
Rationale:

Uncertainty in the clinical and etiological diagnosis of community-acquired pneumonia (CAP) often leads to incorrect treatment and unnecessary use of broad-spectrum antibiotics. Establishing the clinical diagnosis of CAP is hampered by the suboptimal sensitivity of chest radiograph to detect pulmonary infiltrates (~70%). Establishing the etiological diagnosis is also hampered, mainly because of the inevitable diagnostic delays and low sensitivity of routine microbiological tests. There are currently no recommendations for low-dose chest computed tomography (low-dose CT) or viral and bacterial point-of-care multiplex polymerase chain reaction (PoC-PCR) in the diagnostic work-up of CAP patients, because the data supporting such an approach are lacking.

Objective: The aim of this study is to determine the added value of low-dose CT and PoC-PCR in the diagnostic workup of patients with CAP hospitalised to non-intensive care unit (ICU) wards in minimizing selective antibiotic pressure while maintaining patient safety.

Study design: Cluster-randomised controlled trial with historical control period.

Study population: Adult patients (>=18 years old) with a clinical diagnosis of CAP requiring hospitalisation to a non-ICU ward.

Intervention: Intervention arm 1: availability of PoC-PCR during the ER visit; intervention arm 2: performing low-dose CT from the ER or at least within 24 hours; control arm: standard care.

Main study parameters/endpoints: The primary effectiveness outcome is days of therapy of broad-spectrum antibiotics. The primary safety outcome, on which the sample size is calculated, is 90-day all-cause mortality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no risks associated with performing the PoC-PCR and the radiation of the low-dose CT is of negligible risk. Nasopharyngeal swab collection causes a temporary unpleasant sensation. The low-dose CT can reveal unexpected findings which may require additional diagnostic procedures, for which the treating physician will use state-of-the-art guidelines. Treatment recommendations to de-escalate or stop antibiotic treatment may be beneficial for the individual patient by minimising exposure to antibiotics and improve targeted use of antibiotics. Final decisions are always made by the treating physician taking into account all clinical information.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above;
* working diagnosis of CAP at the emergency department with the presence of at least two clinical criteria or one clinical criterion and radiological evidence of CAP, with no other explanation for the signs and symptoms;
* requiring hospitalisation to a non-ICU ward via the ER.

Exclusion Criteria:

* Hospitalisation for two or more days in the last 14 days;
* Residence in a long-term care facility in the last 14 days;
* History of cystic fibrosis;
* Severe immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3555 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Days of therapy of broad-spectrum antibiotics | throughout hospitalization, an average of 7 days
  Days of treatment with broad-spectrum antibiotics during index admission. This will include antibiotic prescriptions provided at discharge.
All-cause mortality | 90 days
  All-cause mortality within 90 days of admission.

SECONDARY OUTCOMES:
days of therapy with any antibiotic | throughout hospitalization, an average of 7 days
  Number of days of treatment with any antibiotics during index admission, including antibiotic prescriptions provided at discharge.
all-cause mortality | 30 days
length of hospital stay | throughout hospitalization, an average of 7 days
adverse outcomes | 90 days
  Composite endpoint comprising ICU admission, in-hospital mortality, and readmission
time to results | throughout hospitalization, an average of 7 days
  Time from admission to availability of the low-dose CT / PoC-PCR results.
time to treatment recommendations | throughout hospitalization, an average of 7 days
  Time from admission to provision of a treatment recommendation following the low-dose CT / PoC-PCR results.
change in antibiotic consumption | throughout hospitalization, an average of 7 days
  Whether changes were made in the antibiotic class during treatment
time to change in antibiotic consumption | throughout hospitalization, an average of 7 days
  When changes were made in the antibiotic class during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marc JM Bonten, MD, PhD, Principal Investigator — University Medical Center Utrecht, the Netherlands
Locations (7):
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Ter Gooi Ziekenhuis, Hilversum
  - University Medical Center, Utrecht
  - Maxima MC, Veldhoven
  - Langeland Ziekenhuis, Zoetermeer

IPD SHARING:
Plan to Share IPD: Undecided